CLINICAL TRIAL: NCT04830241
Title: Neonatal Hypotonia Associated With in Utero Exposure to Antidepressant-Analysis of Two Pharmacovigilance Databases
Brief Title: Neonatal Hypotonia Associated With in Utero Exposure to Antidepressant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: HYPOTONIA
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Neonatal Hypotonia; Antidepressant Drug Adverse Reaction; Pregnancy Related
MeSH Terms: conditions — Muscle Hypotonia | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antidepressant — Cases reported in the World Health Organization (WHO) and the French pharmacovigilance database of neonatal hypotonia newborns following in utero exposure to antidepressant drugs, with a chronology compatible with the drug toxicity
  Other Names: in utero exposure to antidepressant drugs

SUMMARY:
To better characterize the neonatal hypotonia associated with in utero exposure to antidepressants, so far limited to clinical cases, we will perform an observational retrospective pharmacovigilance study, using two databases. First, disproportionality analysis in Vigibase®, the World Health Organization global database, will be perform between antidepressant drugs and neonatal hypotonia . Second, narratives from the French National Pharmacovigilance Database will be extracted.

ELIGIBILITY:
Inclusion Criteria:

* neonatal hypotonia newborns cases associated with in utero exposure to antidepressant drugs

Exclusion Criteria:

* Reports with maternal suicide, congenital malformation and hypotonia occurring only during breastfeeding

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all neonatal hypotonia newborns cases associated with in utero exposure to antidepressant drugs retrived in the two pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
neonatal hypotonia | Case reported in the World Health Organization (WHO) pharmacovigilance database to April 1st 2021
  Identification and extractions of cases of neonatal hypotonia newborns following in utero exposure to antidepressant drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No